CLINICAL TRIAL: NCT02418884
Title: The Impact of Rosuvastatin on the Density Score of Coronary Artery Calcification in CAD Patients With Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Guo Sheng Fu, MD/PhD, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ESR-14-10098
Record Dates: First submitted 2015-03-30; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAD+DM (Other): Using self controlled study to validate the hypothesis that the treatment of rosuvastatin could increase the score of CAC density in CAD patients with diabetes mellitus.
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — CAD patients with diabetes who confirmed CAC will receive rosuvastatin (20mg/d) therapy for 24 months.
  Other Names: Crestor

SUMMARY:
This study is designed to validate the hypothesis that the treatment of rosuvastatin could increase the score of Calcification of Coronary artery(CAC) density in coronary artery disease(CAD) patients with diabetes mellitus.CAD patients with diabetes who confirmed CAC will receive rosuvastatin (20mg/d) therapy for 24 months.

DETAILED DESCRIPTION:
Calcification of atherosclerotic plaque is a complicated and organic active process, which is one of the main pathologic features of atherosclerosis. Widely coverage of CAC is correlated with the greater likelihood of coronary events.With the increasing density of CAC, the risk of cardiovascular disease (CVD) declines.Some studies showed that the calcified plaque in stable CHD is denser.

Statins are widely used in the treatment of atherosclerotic cardiovascular disease. Treatment of statins may increase the density score of CAC, thus, promote the unstable atherosclerotic plaque to the stable plaque.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male and female adults aged 18-70 years old
3. CHD patients without stent implantation determined by coronary angiography or coronary CT examination;
4. Combined with type 2 diabetes: HbA1c≥6.5%, FPG≥7.0mmol/L, 2h blood glucose≥11.1mmol/L
5. Patients who confirmed CAC(Agatston score ≥50,measured by 64 row spiral CT6)

Exclusion Criteria:

1. CHD Patients plan to recieve coronary stenting implantation or coronary artery bypass grafting;
2. Patients combined with severe pulmonary, liver and kidney dysfunction
3. Classed as III-IV grade of New York Heart Association functional
4. Pregnancy test was positive，lactation woman and in women of child-bearing potential not using appropriate contraceptive measures.
5. Life expectancy within 24 months or less
6. Patients combined valvular heart disease and cardiomyopathy
7. Patients combined cancer
8. Patients with atrial fibrillation
9. Patients who is allergic to statins
10. Patients with myopathy
11. Patients with active liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
the Density Score of Coronary Artery Calcification in CAD patients with Diabetes Mellitus | 24 months

SECONDARY OUTCOMES:
the level of serum sclerostin in CAD patients with diabetes mellitus | 24months
the volume score of CAC in CAD patients with diabetes mellitus | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Guosheng Fu, MD/PhD, Principal Investigator — Sir Run Run Shaw Hospital

REFERENCES:
- [Background] Schoenhagen P, Ziada KM, Kapadia SR, Crowe TD, Nissen SE, Tuzcu EM. Extent and direction of arterial remodeling in stable versus unstable coronary syndromes : an intravascular ultrasound study. Circulation. 2000 Feb 15;101(6):598-603. doi: 10.1161/01.cir.101.6.598. PMID 10673250
- [Background] Leber AW, Knez A, White CW, Becker A, von Ziegler F, Muehling O, Becker C, Reiser M, Steinbeck G, Boekstegers P. Composition of coronary atherosclerotic plaques in patients with acute myocardial infarction and stable angina pectoris determined by contrast-enhanced multislice computed tomography. Am J Cardiol. 2003 Mar 15;91(6):714-8. doi: 10.1016/s0002-9149(02)03411-2. No abstract available. PMID 12633805
- [Background] Shemesh J, Apter S, Itzchak Y, Motro M. Coronary calcification compared in patients with acute versus in those with chronic coronary events by using dual-sector spiral CT. Radiology. 2003 Feb;226(2):483-8. doi: 10.1148/radiol.2262011903. PMID 12563143
- [Background] Ehara S, Kobayashi Y, Yoshiyama M, Shimada K, Shimada Y, Fukuda D, Nakamura Y, Yamashita H, Yamagishi H, Takeuchi K, Naruko T, Haze K, Becker AE, Yoshikawa J, Ueda M. Spotty calcification typifies the culprit plaque in patients with acute myocardial infarction: an intravascular ultrasound study. Circulation. 2004 Nov 30;110(22):3424-9. doi: 10.1161/01.CIR.0000148131.41425.E9. Epub 2004 Nov 22. PMID 15557374
- [Background] Houslay ES, Cowell SJ, Prescott RJ, Reid J, Burton J, Northridge DB, Boon NA, Newby DE; Scottish Aortic Stenosis and Lipid Lowering Therapy, Impact on Regression trial Investigators. Progressive coronary calcification despite intensive lipid-lowering treatment: a randomised controlled trial. Heart. 2006 Sep;92(9):1207-12. doi: 10.1136/hrt.2005.080929. Epub 2006 Jan 31. PMID 16449511
- [Background] Terry JG, Carr JJ, Kouba EO, Davis DH, Menon L, Bender K, Chandler ET, Morgan T, Crouse JR 3rd. Effect of simvastatin (80 mg) on coronary and abdominal aortic arterial calcium (from the coronary artery calcification treatment with zocor [CATZ] study). Am J Cardiol. 2007 Jun 15;99(12):1714-7. doi: 10.1016/j.amjcard.2007.01.060. Epub 2007 Apr 26. PMID 17560880
- [Background] Criqui MH, Denenberg JO, Ix JH, McClelland RL, Wassel CL, Rifkin DE, Carr JJ, Budoff MJ, Allison MA. Calcium density of coronary artery plaque and risk of incident cardiovascular events. JAMA. 2014 Jan 15;311(3):271-8. doi: 10.1001/jama.2013.282535. PMID 24247483
- [Background] Koos R, Brandenburg V, Mahnken AH, Schneider R, Dohmen G, Autschbach R, Marx N, Kramann R. Sclerostin as a potential novel biomarker for aortic valve calcification: an in-vivo and ex-vivo study. J Heart Valve Dis. 2013 May;22(3):317-25. PMID 24151757
- [Background] Brandenburg VM, Kramann R, Koos R, Kruger T, Schurgers L, Muhlenbruch G, Hubner S, Gladziwa U, Drechsler C, Ketteler M. Relationship between sclerostin and cardiovascular calcification in hemodialysis patients: a cross-sectional study. BMC Nephrol. 2013 Oct 10;14:219. doi: 10.1186/1471-2369-14-219. PMID 24112318
- [Derived] Zhang W, Luan Y, Jin C, Xu S, Bi X, Zhao Y, Qiu F, Fu G, Wang M. The Impact of Rosuvastatin on the Density Score of Coronary Artery Calcification in Coronary Artery Disease Patients with Type 2 Diabetes Mellitus: Rationale and Design of RosCal Study. Clin Drug Investig. 2016 Dec;36(12):1023-1029. doi: 10.1007/s40261-016-0445-4. PMID 27541380